CLINICAL TRIAL: NCT01489332
Title: Induction Chemotherapy, Preoperative Radiochemotherapy, Consolidation Chemotherapy, Operation and Adjuvant Chemotherapy in the Treatment of Locally Advanced Rectal Cancer- OIGIT 5-01 Phase II Trial
Brief Title: Induction Chemotherapy,Radiochemotherapy, Consolidation Chemotherapy in Preoperative Treatment of Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 163/06/11
Record Dates: First submitted 2011-11-11; First posted 2011-12-09 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; capecitabine; radiotherapy; locally advanced rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: intensified preoperative chemotherapy — capecitabine 1250 mg/m² p.o. twice daily for 14 consecutive days, 7 days rest for one cycle; radiotherapy: 50.4 Gy to the pelvis (25x 1.8 Gy on days 1-33, excluding weekends) plus 5.4 Gy on days 36-38 as a boost to the primary tumour (3 fractions of 1.8 Gy).Three- dimensional CT planing and a four field box technique with high energy photons (15 MV) will be used. capecitabine 825 mg/m² p.o. twice daily on days 1-38 (including weekends), One week after completion of radiochemotherapy patients receive 2 cycles of capecitabine based chemotherapy (1250 mg/m² p.o. twice daily for 14 consecutive days every three weeks).
  Radical surgery (TME): to be undertaken 8 weeks following completion of chemoradiation Postoperative treatment:capecitabine 1250 mg/m² p.o. twice daily for 14 consecutive days every three weeks; 3 cycles (R0 beginning 6-8 weeks after surgery

SUMMARY:
The use of capecitabine based preoperative chemoradiation and adjuvant chemotherapy is standard treatment of locally advanced rectal cancer. It has reduced local recurrence rate to less than 10%, but has only had limited effect on overall survival due to the constantly high (more than 30%) rate of distant metastasis.

Complete eradication of the primary tumour observed in the histopathological specimen (pathological complete response, pCR) correlates with a favourable overall prognosis so obtaining a pCR might be beneficial. The aim of the study is to investigate whether the addition of capecitabine based chemotherapy before preoperative chemoradiation and also before the operation improves pathological complete remission rate in locally advanced rectal cancer with acceptable toxicity. Secondary objectives are to evaluate pathological downstaging rate, histopathological R0 resection rate,sphincter preservation rate, perioperative surgical complication rate, local control, DFS, OS, late toxicity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with histologically proven adenocarcinoma of the rectum (tumour located below the peritoneum),
* T3/4 or any node positive disease (clinical stage according the TNM classification system)
* No evidence of metastatic disease.
* The disease must be considered either resectable at the time of entry or thought to become resectable after preoperative chemoradiation.
* Age 18 years and more
* WHO Performance Status 0-2
* No prior radiotherapy, chemotherapy or any targeting therapy for rectal cancer
* Adequate hematological, hepatic and renal function Ability to swallow tablets
* Signed informed consent
* Patients must be willing and able to comply with the protocol for duration of the study

Exclusion Criteria:

* Malignancy of the rectum other than adenocarcinoma
* Any unrested synchronous colon cancer
* Other co-existing malignancy or malignancy within the past 5 years, with the exception of adequately treated in situ carcinoma of the cervix or basal cell carcinoma of the skin
* Significant heart disease (uncontrolled hypertension despite of medication (> 150/100 mmHg), NYHA class III or IV heart disease,unstable angina or myocardial infarction within the past 1 year prior the study entry, history of significant ventricular arrhythmia requiring treatment)
* Pregnant or lactating patient
* Females with a positive or no pregnancy test unless childbearing potential can be otherwise excluded (amenorrheic for at least 2 years,hysterectomy or oophorectomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission rate (pCR) | after the pathological examination of surgical speciments ie within 14 days after the operation

SECONDARY OUTCOMES:
Toxicity | According to NCI-CTC (version 3.0): every week for 16 week preoperative, perioperative (0-30 days postoperative), early (30 days - 6 months postoperative), and late (more than 6 months postoperative)
  Number of patients with adverse events and the grade of adverse events
Histopathological R0 resection rate | after the pathological examination of resected speciments ie within 14 days after the operation
Loco-regional failure rate | after 3y and 5y of operation
Disease-free survival | after 3y and 5y of operation
Overall survival | after 3y and 5y of the operation
Quality of life | before the treatment, after 1,and 3 years of the operation
  We will use EORTC questionnaires QLQ C30 and C38

CONTACTS AND LOCATIONS:
Overall Officials: Vaneja Velenik, Prof.assist, Principal Investigator — Institute of Oncology Ljubljana, Slovenia
Locations (1):
- Institute of Oncology, Ljubljana, Slovenia

REFERENCES:
- [Background] Habr-Gama A, Perez RO, Nadalin W, Sabbaga J, Ribeiro U Jr, Silva e Sousa AH Jr, Campos FG, Kiss DR, Gama-Rodrigues J. Operative versus nonoperative treatment for stage 0 distal rectal cancer following chemoradiation therapy: long-term results. Ann Surg. 2004 Oct;240(4):711-7; discussion 717-8. doi: 10.1097/01.sla.0000141194.27992.32. PMID 15383798
- [Background] Velenik V, Oblak I, Anderluh F. Long-term results from a randomized phase II trial of neoadjuvant combined-modality therapy for locally advanced rectal cancer. Radiat Oncol. 2010 Sep 29;5:88. doi: 10.1186/1748-717X-5-88. PMID 20920276
- [Background] Ruo L, Tickoo S, Klimstra DS, Minsky BD, Saltz L, Mazumdar M, Paty PB, Wong WD, Larson SM, Cohen AM, Guillem JG. Long-term prognostic significance of extent of rectal cancer response to preoperative radiation and chemotherapy. Ann Surg. 2002 Jul;236(1):75-81. doi: 10.1097/00000658-200207000-00012. PMID 12131088
- [Background] Bujko K, Glynne-Jones R, Bujko M. Adjuvant chemotherapy for rectal cancer. Ann Oncol. 2010 Dec;21(12):2443. doi: 10.1093/annonc/mdq616. No abstract available. PMID 21098619
- [Background] Bujko K, Glynne-Jones R, Bujko M. Does adjuvant fluoropyrimidine-based chemotherapy provide a benefit for patients with resected rectal cancer who have already received neoadjuvant radiochemotherapy? A systematic review of randomised trials. Ann Oncol. 2010 Sep;21(9):1743-1750. doi: 10.1093/annonc/mdq054. Epub 2010 Mar 15. PMID 20231300
- [Background] Habr-Gama A, Perez RO, Sabbaga J, Nadalin W, Sao Juliao GP, Gama-Rodrigues J. Increasing the rates of complete response to neoadjuvant chemoradiotherapy for distal rectal cancer: results of a prospective study using additional chemotherapy during the resting period. Dis Colon Rectum. 2009 Dec;52(12):1927-34. doi: 10.1007/DCR.0b013e3181ba14ed. PMID 19934911